CLINICAL TRIAL: NCT06249815
Title: Sequential Use of Foley's Catheter and Low Dose Oral Misoprostol Versus Misoprostol Alone for Induction of Labour : a Multicentre Randomised Controlled Trial
Brief Title: Sequential Use of Foley's Catheter and Misoprostol Versus Misoprostol Alone for Induction of Labour: a Multicentre Randomised Controlled Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kazakhstan's Medical University "KSPH" (Other)
Collaborators: Asfendiyarov Kazakh National Medical University (Other)
Responsible Party: Principal Investigator, Dilfuza Sultanmuratova, principal investigator, Kazakhstan's Medical University "KSPH"
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-23-2024
Record Dates: First submitted 2024-01-12; First posted 2024-02-08 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Induction of Labor
Keywords: Induction of labor; low dose misoprostol; Foley Catheter
MeSH Terms: interventions — Misoprostol; Silicones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Foley catheter + misoprostol (Active Comparator): -cervical ripening with transcervical Foley catheter 22 F for 16 hours, then sequentially 25 μg oral misoprostol once every 2 hour.Max 200 μg
  Interventions: Combination Product: Misoprostol 200mcg Tab
- misoprostol (Active Comparator): 25 μg oral misoprostol alone once every 2 hour, Max 200 μg.
  Interventions: Drug: Misoprostol 200mcg Tab

INTERVENTIONS:
Combination Product: Misoprostol 200mcg Tab — ranscervical Foley catheter (silicone, size 20F with 30ml balloon)+Misoprostol 200 mcg dissolvedwith 200 ml water and divided to 25ml solution every 2 hours per os for maximum of 8 doses
  Other Names: Transcervical Foley catheter (silicone, size 20F with 30ml balloon)
  Arms: Foley catheter + misoprostol
Drug: Misoprostol 200mcg Tab — Misoprostol 200 mcg dissolvedwith 200 ml water and divided to 25ml solution every 2 hours per os for maximum of 8 doses
  Arms: misoprostol

SUMMARY:
Evaluation of efficacy of inducing labour using a Foley's catheter and low dose oral misoprostol sequentially, in comparison with low dose oral misoprostol alone.

DETAILED DESCRIPTION:
a multicentre, open-label randomised controlled trial in 2 hospitals in the Almaty,Kazakhstan. Women with a term singleton pregnancy in cephalic presentation, an unfavourable cervix, intact membranes, and without a previous caesarean section will be randomly allocated to 2 groups: 1 group -cervical ripening with Foley's catheter for 16 hour and sequentially 25 μg oral misoprostol once every 2 hour, 2 nd group- 25 μg oral misoprostol once every 2 hour. The primary outcome will be vaginal delivery within 24 hours(to evaluate effectiveness) and secondary outcoms 1-5-min Apgar score and hospitalization in ICU, rate of hyperstimulation ,hemorrage,chorioamnionitis (for evaluating safety)

ELIGIBILITY:
Inclusion Criteria:

* women with an unfavourable cervix who will scheduled for induction of labour

Exclusion Criteria:

* Women with previous caesarean sections unable to give informed consent Multiple pregnancy History of allergy to misoprostol Ruptured membranes All cases when physiological childbirth is impossible (placenta previa,transverse position of the fetus )

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2024-04-26 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Efficiency of induction | 24 hours.
  Number of Participants with vaginal births

SECONDARY OUTCOMES:
Safety for baby | 5 minutes
  Rate of cases Apgar score <7 points
Safety for mother | 24 hour
  incidence of hyperstimulation
rete of hemorrage | 24 hour
  bleeding more than 500 ml during the vaginal delivery, more than 1000 ml after c-section
rate of chorioamnionitis chorioamnionitis | 24 hour
  meconial amniotic fluid, tachycardia, leukocytosis

CONTACTS AND LOCATIONS:
Overall Officials: Saule Issenova, Study Chair — Asfendiyarov Kazakh National Univercity; DILFUZA SULTANMURATOVA, Principal Investigator — Kazakhstans Medical Uivercity
Locations (2):
- Kazakhstan (2):
  - City Perinatology Centre 3, Almaty
  - Center for Perinatology and Pediatric Cardiac Surgery, Almaty

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR